CLINICAL TRIAL: NCT02097641
Title: Prospective, Randomized, Multi-center Phase 2 Clinical Trial of Allogeneic Bone Marrow-derived Human Mesenchymal Stromal Cells (hMSCs) for the Treatment of Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Human Mesenchymal Stromal Cells For Acute Respiratory Distress Syndrome (START)
Acronym: START
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael A. Matthay (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts General Hospital (Other); Stanford University (Other); University of Pittsburgh (Other); University of Minnesota (Other); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Michael A. Matthay, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSF-hMSC-ARDS-P2; 1U01HL108713-01 (NIH)
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Allogeneic Bone Marrow-derived Human Mesenchymal Stromal Cells; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Mesenchymal Stromal Cells (hMSCs) (Experimental): A single dose of 10 million cells/kg PBW (predicted body weight) Allogeneic Bone Marrow-Derived Human Mesenchymal Stromal Cells was administered intravenously over approximately 60-80 minutes.
  Interventions: Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stromal Cells
- Plasma-Lyte A (placebo) (Placebo Comparator): A single dose of Plasma-Lyte A was administered intravenously over approximately 60-80 minutes.
  Interventions: Biological: Plasma-Lyte A

INTERVENTIONS:
Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stromal Cells — Allogeneic Bone Marrow-Derived Human Mesenchymal Stromal Cells was administered intravenously over approximately 60-80 minutes.
  Arms: Human Mesenchymal Stromal Cells (hMSCs)
Biological: Plasma-Lyte A — Plasma-Lyte A placebo was administered intravenously over approximately 60-80 minutes.
  Arms: Plasma-Lyte A (placebo)

SUMMARY:
This was a Phase 2a, randomized, double-blind, placebo-controlled, multi-center trial to assess the safety and efficacy of a single dose of Allogeneic Bone Marrow-derived Human Mesenchymal Stromal Cells (hMSCs) infusion in patients with Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
We carried out a randomized, double-blind placebo-controlled trial of allogeneic bone marrow derived human mesenchymal stromal cells for treatment of moderate to severe ARDS in 60 patients, 40 MSC and 20 placebo, in a 2:1 randomization. This trial is the extension of the Phase 1 pilot trial (NCT01775774). Patients were followed daily for adverse events through day 28, death or hospital discharge, whichever occurs first. Vital status was collected at 6 and 12 months after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they meet all of the below criteria. Criteria 1-3 must all be present within a 24-hour time period and at the time of enrollment:

Acute onset (defined below) of:

1. A need for positive pressure ventilation by an endotracheal or tracheal tube with a PaO2/FiO2 ratio < 200 with at least 8 cm H2O positive end-expiratory airway pressure (PEEP)
2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph
3. No clinical evidence of left atrial hypertension for bilateral pulmonary infiltrates.

Exclusion Criteria:

1. Age less than 18 years
2. Greater than 96 hours since first meeting ARDS criteria per the Berlin definition of ARDS
3. Pregnant or breast-feeding
4. Prisoner
5. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last 2 years
6. Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
7. Moderate to severe liver failure (Childs-Pugh Score > 12)
8. Severe chronic respiratory disease with a PaCO2 > 50 mm Hg or the use of home oxygen
9. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
10. Major trauma in the prior 5 days
11. Lung transplant patient
12. No consent/inability to obtain consent
13. Moribund patient not expected to survive 24 hours
14. World Health Organization (WHO) Class III or IV pulmonary hypertension
15. Documented deep venous thrombosis or pulmonary embolism within past 3 months
16. No arterial line/no intent to place an arterial line
17. No intent/unwillingness to follow lung protective ventilation strategy or fluid management protocol
18. Currently receiving extracorporeal life support (ECLS) or high-frequency oscillatory ventilation (HFOV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Matthay, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Saint Paul, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matthay MA, Calfee CS, Zhuo H, Thompson BT, Wilson JG, Levitt JE, Rogers AJ, Gotts JE, Wiener-Kronish JP, Bajwa EK, Donahoe MP, McVerry BJ, Ortiz LA, Exline M, Christman JW, Abbott J, Delucchi KL, Caballero L, McMillan M, McKenna DH, Liu KD. Treatment with allogeneic mesenchymal stromal cells for moderate to severe acute respiratory distress syndrome (START study): a randomised phase 2a safety trial. Lancet Respir Med. 2019 Feb;7(2):154-162. doi: 10.1016/S2213-2600(18)30418-1. Epub 2018 Nov 16. PMID 30455077
- [Derived] Wick KD, Leligdowicz A, Zhuo H, Ware LB, Matthay MA. Mesenchymal stromal cells reduce evidence of lung injury in patients with ARDS. JCI Insight. 2021 Jun 22;6(12):e148983. doi: 10.1172/jci.insight.148983. PMID 33974564
- [Derived] Liu KD, Wilson JG, Zhuo H, Caballero L, McMillan ML, Fang X, Cosgrove K, Calfee CS, Lee JW, Kangelaris KN, Gotts JE, Rogers AJ, Levitt JE, Wiener-Kronish JP, Delucchi KL, Leavitt AD, McKenna DH, Thompson BT, Matthay MA. Design and implementation of the START (STem cells for ARDS Treatment) trial, a phase 1/2 trial of human mesenchymal stem/stromal cells for the treatment of moderate-severe acute respiratory distress syndrome. Ann Intensive Care. 2014 Jul 3;4:22. doi: 10.1186/s13613-014-0022-z. eCollection 2014. PMID 25593740
- [Derived] Asmussen S, Ito H, Traber DL, Lee JW, Cox RA, Hawkins HK, McAuley DF, McKenna DH, Traber LD, Zhuo H, Wilson J, Herndon DN, Prough DS, Liu KD, Matthay MA, Enkhbaatar P. Human mesenchymal stem cells reduce the severity of acute lung injury in a sheep model of bacterial pneumonia. Thorax. 2014 Sep;69(9):819-25. doi: 10.1136/thoraxjnl-2013-204980. Epub 2014 Jun 2. PMID 24891325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 24, 2014, to Feb 9, 2017, 1038 patients were screened for eligibility, of whom 975 were excluded, and 63 were randomly assigned to a treatment group. Three patients were not eligible for treatment after randomization and, therefore, 40 patients received human mesenchymal stem cells and 20 patients received placebo.
Pre-assignment Details: Three patients who were randomly assigned to receive human mesenchymal stem cells, were excluded: 2 did not meet baseline stability criteria; 1 patient's PaO2:FiO2 > 200 mmHg.
Groups:
- Human Mesenchymal Stem Cells: A single dose of 10 million cells/kg PBW (predicted body weight) Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells administered intravenously over approximately 60-80 minutes.
  Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells will be administered intravenously over approximately 60-80 minutes.
- Plasma-Lyte A: A single dose of Plasma-Lyte A will be administered intravenously over approximately 60-80 minutes.
  Plasma-Lyte A: Plasma-Lyte A placebo will be administered intravenously over approximately 60-80 minutes.
Period: Overall Study
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Human Mesenchymal Stem Cells (hMSCs): A single dose of 10 million cells/kg PBW (predicted body weight) Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells administered intravenously over approximately 60-80 minutes.
  Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells will be administered intravenously over approximately 60-80 minutes.
- Plasma-Lyte A (Placebo): A single dose of Plasma-Lyte A will be administered intravenously over approximately 60-80 minutes.
  Plasma-Lyte A: Plasma-Lyte A placebo will be administered intravenously over approximately 60-80 minutes.
- Total: Total of all reporting groups
Arm/Group | Human Mesenchymal Stem Cells (hMSCs) | Plasma-Lyte A (Placebo) | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 12 | 42
  >=65 years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (17) | 55 (20) | 55 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 31 | 16 | 47
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 4 | 1 | 5
  White | 27 | 13 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60
Cause of Acute Respiratory Distress Syndrome (ARDS) [Count of Participants; unit: Participants]
  Sepsis with pneumonia | 19 | 12 | 31
  Sepsis without pneumonia | 5 | 2 | 7
  Pneumonia without sepsis | 11 | 5 | 16
  Aspiration only | 4 | 1 | 5
  Other | 1 | 0 | 1
Arterial pressure [Mean (Standard Deviation); unit: mm Hg] | 75 (10) | 76 (9) | 75 (10)
Taking vasopressors at the time of infusion [Count of Participants; unit: Participants] | 24 | 9 | 33
Sequential Organ Failure Assessment (SOFA) [Mean (Standard Deviation); unit: units on a scale] — SOFA score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems which are added up. Each score ranges from 0 to 4. SOFA score ranges from 0 (best) to 24 (worst). Population: Data not recorded in one patient treated with Plasma-Lyte A (placebo).
  units on a scale
    number analyzed (Participants) | 40 | 19 | 59
    (all) | 8.1 (3.3) | 6.9 (2.7) | 7.7 (3.2)
Acute Physiologic Assessment and Chronic Health Evaluation (APACHE) III score [Mean (Standard Deviation); unit: units on a scale] — The range of APACHE III is from 0 to 299. The higher score, the worse clinical outcome. Population: Data not recorded in one patient treated with Plasma-Lyte (placebo).
  units on a scale
    number analyzed (Participants) | 40 | 19 | 59
    (all) | 104 (31) | 89 (33) | 99 (32)
Minute ventilation [Mean (Standard Deviation); unit: L/min] | 11.1 (3.2) | 9.6 (2.4) | 10.6 (3.0)
Respiratory rate [Mean (Standard Deviation); unit: breaths/min] | 27.8 (6.6) | 24.5 (6.3) | 26.7 (6.6)
Tidal volume [Mean (Standard Deviation); unit: mL/kg predicted body weight] — Population: Data not recorded in one patient treated with hMSCs.
  mL/kg predicted body weight
    number analyzed (Participants) | 39 | 20 | 59
    (all) | 6.3 (0.9) | 6.1 (0.7) | 6.2 (0.9)
Mean airway pressure [Mean (Standard Deviation); unit: cm H2O] — Population: Data not recorded in three patients treated with hMSCs and one patient treated with Plasma-Lyte A (placebo).
  cm H2O
    number analyzed (Participants) | 37 | 19 | 56
    (all) | 17.8 (4.9) | 16.4 (3.6) | 17.4 (4.6)
Plateau airway pressure [Mean (Standard Deviation); unit: cm H2O] — Population: 15 patients did not have baseline plateau pressure recorded.
  cm H2O
    number analyzed (Participants) | 30 | 15 | 45
    (all) | 26.4 (5.7) | 23.7 (5.1) | 25.5 (5.6)
Positive end-expiratory pressure (PEEP) [Mean (Standard Deviation); unit: cm H2O] | 12.4 (3.7) | 10.8 (2.6) | 11.8 (3.4)
Driving pressure [Mean (Standard Deviation); unit: cm H2O] — Population: Data not recorded in 10 patients treated with hMSCs and in 5 patients treated with Plasma-Lyte (placebo).
  cm H2O
    number analyzed (Participants) | 30 | 15 | 45
    (all) | 14.0 (4.1) | 12.5 (4.3) | 13.5 (4.2)
PaO2/FiO2 [Mean (Standard Deviation); unit: kPa] | 18.1 (4.3) | 19.1 (5.2) | 18.4 (4.6)
Oxygenation index [Mean (Standard Deviation); unit: kPa] — Oxygenation index calculated as: FiO2 (%) x Mean Airway Pressure / PaO2 Population: Data not recorded in 3 patients treated with hMSCs and 1 patient treated with Plasma-Lyte (placebo).
  kPa
    number analyzed (Participants) | 37 | 19 | 56
    (all) | 108.1 (45.9) | 95.7 (41.2) | 103.9 (44.4)
Lung injury score (LIS) [Mean (Standard Deviation); unit: units on a scale] — LIS is a composite 4-point scoring system including the PaO2/FiO2, PEEP, lung compliance, and the extent of infiltrates on the chest X-ray. Each of the four components is categorized from 0 to 4, where a higher number is worse. The total Lung Injury Score is obtained by dividing the aggregate sum by the number of components used.
  units on a scale | 3.1 (0.4) | 3.0 (0.5) | 3.1 (0.4)
Ventilation mode [Count of Participants; unit: Participants]
  Volume control | 37 | 17 | 54
  Pressure-regulated volume control | 1 | 2 | 3
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Patients Occurred Pre-specified Infusion Associated Events Occurring Within 6 Hours of Study Infusion
Description: Within 6 h of study product infusion:
  * Increase in vasopressor dose to the following values or higher:
  * Norepinephrine 10 μg/min
  * Phenylephrine 100 μg/min
  * Dopamine 10 μg/kg per min
  * Epinephrine 0.1 μg/kg per min or addition of a third vasopressor
  * New ventricular tachycardia, ventricular fibrillation or asystole
  * New cardiac arrhythmia requiring cardioversion
  * Hypoxaemia requiring an increase in FiO2 of 0·2 or more and an increase in PEEP of 5·0 or more to maintain SpO2 in the target range of 88-95%
  * Clinical scenario consistent with transfusion incompatibility or transfusion-related infection (eg, urticaria, new bronchospasm)
Time Frame: 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stem Cells (hMSCs) | Plasma-Lyte A (Placebo)
Number analyzed (Participants) | 40 | 20
Participants | 0 | 0

2. Primary Outcome: Numbers of Patients Occurred Any Cardiac Arrest or Death Within 24 Hours of Study Infusion
Description: Within 24 h of study product infusion
  • Any cardiac arrest or death
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stem Cells (hMSCs) | Plasma-Lyte A (Placebo)
Number analyzed (Participants) | 40 | 20
Participants | 1 | 0

3. Primary Outcome: Numbers of Patients Occurred Any Unexpected Severe Adverse Events (Including All-cause Deaths)
Description: Safety endpoint: Any unexpected severe adverse events in two groups
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 40 | 20
Participants | 20 | 5

4. Secondary Outcome: PaO2:FiO2 Change From Baseline to Day 3
Description: Efficacy endpoint: PaO2:FiO2 change from baseline to day 3
Time Frame: baseline and day 3
Population: The values of PaO2:FiO2 were not available in 10 patients treated with hMSCs and in 2 patients treated with placebo.
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 30 | 18
kPa | 3.7 [-1.2 to 10.8] | 3.5 [-2.7 to 8.3]

5. Secondary Outcome: Lung Injury Score From Baseline to Day 3
Description: Murray score for acute lung injury. The range is 0 to 4. The higher score, the worst outcome.
Time Frame: baseline and day 3
Population: The values were missing in 9 hMSC patients and 2 placebo patients.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 31 | 18
units on a scale | -0.50 [-1.00 to -0.25] | -0.33 [-0.67 to -0.08]

6. Secondary Outcome: Oxygenation Index Change From Baseline to Day 2
Description: Oxygenation index with the following validated measure of respiratory function: FiO2 (%) x mean airway pressure / PaO2
Time Frame: baseline and day 2
Population: The values were missing in 16 patients treated by MSC and 6 patients treated by placebo
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 24 | 14
kPa | -30.3 [-67.9 to 14.9] | -19.5 [-47.8 to 10.9]

7. Secondary Outcome: SOFA Score Change From Baseline to Day 3
Description: Sequential organ failure assessment score (SOFA). The SOFA score ranges from 0 to 24. The higher, the worse.
Time Frame: baseline and day 3
Population: The values were missing in 3 MSC patients and 1 placebo patient.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 37 | 19
units on a scale | -2 [-4 to 0] | -1 [-4 to 1]

8. Secondary Outcome: Number of Patients Death to Day 28
Description: Efficacy endpoint: all-cause mortality at day 28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 40 | 20
Participants | 12 | 3

9. Secondary Outcome: Mortality to Day 60
Description: Efficacy endpoint: all-cause mortality at day 60
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 40 | 20
Participants | 15 | 5

10. Secondary Outcome: Number of Ventilator-free Days to Day 28
Description: Efficacy endpoint: Number of ventilator-free days to day 28.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 40 | 20
days | 2 [0 to 23] | 17 [0 to 24]

11. Secondary Outcome: Non-pulmonary Organ-failure-free Days to Day 28
Description: Efficacy endpoint: Non-pulmonary organ-failure-free days to day 28
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 40 | 20
days | 12 [4 to 24] | 8 [4 to 15]

12. Secondary Outcome: Angiopoietin 2 Change From Baseline to 6 h
Description: Biological markers of endothelial injury: angiopoietin 2
Time Frame: baseline and 6 hours
Population: The biomarker values were missing in one patient treated with hMSC and one patient treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 39 | 19
pg/mL | -1120 [-4706 to -66] | 287 [-1005 to 2374]

13. Secondary Outcome: Angiopoietin 2 Change From Baseline to 24 h
Description: Biological markers of endothelial injury: angiopoietin 2
Time Frame: baseline and 24 hours
Population: The values were not available in two patients treated with hMSC and two patients treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 38 | 18
pg/mL | -2080 [-6404 to 47] | -537 [-4294 to 1029]

14. Secondary Outcome: Interleukin 6 Change From Baseline to 6 h
Description: Biological markers of inflammation: interleukin 6
Time Frame: baseline and 6 hours
Population: The values were not available in one patient treated with hMSC and one patient treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 39 | 19
pg/mL | -51 [-124 to 4] | -20 [-71 to 17]

15. Secondary Outcome: Interleukin 6 Change From Baseline to 24 h
Description: Biological markers of inflammation: interleukin 6
Time Frame: baseline and 24 hours
Population: The values were not available in two patients treated with hMSC and two patients treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 38 | 18
pg/mL | -34 [-137 to 4] | -43 [-165 to 39]

16. Secondary Outcome: Interleukin 8 Change From Baseline to 6 h
Description: Biological markers of inflammation: interleukin 8
Time Frame: baseline and 6 hours
Population: The values were not available in one patient treated with hMSC and one patient treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 39 | 19
pg/mL | -2 [-24 to 3] | -1 [-8 to 1]

17. Secondary Outcome: Interleukin 8 Change From Baseline to 24 h
Description: Biological markers of inflammation: interleukin 8
Time Frame: baseline and 24 hours
Population: The values were not available in two patients treated with hMSC and two patients treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 38 | 18
pg/mL | -5 [-34 to 4] | -5 [-17 to -1]

18. Secondary Outcome: RAGE Change From Baseline to 6 h
Description: Biological markers of alveolar epithelial injury: receptor for advanced glycation end products (RAGE)
Time Frame: baseline and 6 hours
Population: The values were not available in one patient treated with hMSC and one patient treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 39 | 19
pg/mL | -326 [-888 to -45] | -322 [-624 to -93]

19. Secondary Outcome: RAGE Change From Baseline to 24 h
Description: Biological markers of alveolar epithelial injury: receptor for advanced glycation end products (RAGE)
Time Frame: baseline and 24 hours
Population: The values were not available in two patients treated with hMSC and two patients treated with placebo.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
Number analyzed (Participants) | 38 | 18
pg/mL | -393 [-1118 to -78] | -411 [-1057 to -110]

ADVERSE EVENTS:
Time Frame: 60 days
Description: 1. All-cause mortality by day 60 after study product infusion
  2. Serious adverse events, expected and unexpected, also included any deaths through study day 28 (none of them were related to study product or study procedures per DSMB review)
  3. Please see our Lancet Resp Medicine 2018 publication (citation included) for further details including adjusted analyses of baseline differences between the MSC and placebo treated groups
Arm/Group | Human Mesenchymal Stem Cells | Plasma-Lyte A
All-Cause Mortality (participants affected / at risk) | 15/40 | 5/20
Serious Adverse Events (participants affected / at risk) | 17/40 | 11/20
Other Adverse Events (participants affected / at risk) | 2/40 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human Mesenchymal Stem Cells (N=40) | Plasma-Lyte A (N=20)
Lower extremity weakness (Nervous system disorders) | 0 (0) | 1 (1)
Hospital readmission due to post-surgical pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospital readmission due to pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diffuse alveolar hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death due to cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Heart block (Cardiac disorders) | 1 (1) | 0 (0)
Ischemic stroke (Cardiac disorders) | 0 (0) | 1 (1)
Liver abscess (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute pancreatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death due to worsening respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Worsening respiratory failure, recovered (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Calvarial bone marrow abnormality (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Death due to multi-organ failure (General disorders) | 8 (8) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Human Mesenchymal Stem Cells (N=40) | Plasma-Lyte A (N=20)
Hepatitis (Hepatobiliary disorders) | 1 | 0
Fecal and urinary incontinence (Renal and urinary disorders) | 0 | 1
Deep venous thrombosis (Vascular disorders) | 1 | 0
Acute anemia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02097641/Prot_SAP_000.pdf